CLINICAL TRIAL: NCT07375225
Title: Evaluation of Adherence, Persistence and Efficacy of Treatment With Alirocumab 300mg in Italy - The ALINET Registry
Brief Title: Evaluation of Adherence, Persistence and Efficacy of Treatment With Alirocumab 300mg in Italy
Acronym: ALINET
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: Prot. 28/2024
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with hyperlipidaemia under Alirocumab 300 mg treatment.: Subjects with hyperlipidaemia
  Interventions: Drug: Praluent (Alirocumab)

INTERVENTIONS:
Drug: Praluent (Alirocumab) — Alirocumab 300 mg injection

SUMMARY:
Evaluation of adherence, persistence and efficacy of treatment with alirocumab 300 mg in a real-life Italian population.

ELIGIBILITY:
Inclusion Criteria:

- Patients under alirocumab 300mg treatment.

Exclusion Criteria:

* Age < 18 years o > 80 years;
* Patients who refuse to participate and to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients from Italy, who have received alirocumab 300mg as part of routine clinical management of their hyperlipidaemia at time of enrollment, based on national reimbursement criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Description of adherence of treatment with alirocumab 300mg in a real-life Italian population. | 6-12-24-36 months
  Adherence will be assessed in terms of Medical Possession Ratio (MPR) which is defined as the ratio between the treatment units dispensed during the treatment period and the duration of the treatment period itself.
Description of persistence of treatment with alirocumab 300mg in a real-life Italian population. | 6-12-24-36 months
  Persistence will be assessed in terms of therapeutic continuity from the start of treatment to enrollment.
Description of efficacy of treatment with alirocumab 300mg in a real-life Italian population. | 6-12-24-36 months
  Efficacy of treatment will be evaluated as a change in the LDL (deltaLDL) value from the start of treatment (percentage and absolute value).

SECONDARY OUTCOMES:
Description of safety of treatment with alirocumab 300mg in a real-life Italian population. | 6-12-24-36 months
  Safety will be evaluated in terms of adverse reactions or intolerance to the drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli, Napoli, Italy